CLINICAL TRIAL: NCT04159714
Title: Bandage Contact Lens Application for the Management of Corneal Abrasion in the Emergency Department
Brief Title: Bandage Contact Lens Application for the Management of Corneal Abrasion
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in practice decreasing availability of eligible patients.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Robert J. Hyde, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-009586
Record Dates: First submitted 2019-11-08; First posted 2019-11-12 (Actual); Results first posted 2023-01-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2022-12

CONDITIONS: Corneal Abrasion
MeSH Terms: conditions — Corneal Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Bandage Contact Lens (BCL) group (Experimental): Subjects diagnosed with superficial corneal abrasion in the Emergency Department will have a bandage contact lens soaked in antibiotic solution placed in the affected eye
  Interventions: Device: Air Optix contact lens
- Usual Care Group (No Intervention): Subjects diagnosed with superficial corneal abrasion in the Emergency Department will have usual care provided in the Emergency Department

INTERVENTIONS:
Device: Air Optix contact lens — Contact lens will be placed on the surface of the patient's eye and is to be used as a bandage
  Arms: Bandage Contact Lens (BCL) group

SUMMARY:
The researchers are trying to understand if the application of a bandage contact lens results in better relief than usual treatment for a corneal abrasion.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Superficial Corneal Abrasion

Exclusion Criteria:

* Incarceration
* Pregnancy
* Inability to Provide Informed Consent
* Infectious keratitis
* Retained foreign bodies in the eye
* Active infection involving the orbit or periorbital region
* Patients who are not able to or who are deemed unlikely to follow-up with ophthalmology
* A history or recent contact lens wear
* A lack of trauma or an unclear history of trauma as the inciting cause of the abrasion
* Allergy to the antimicrobial solution (POLYTRIM)
* Women who are currently breastfeeding
* Chronic eye drop use
* A history of eye surgery other than cataract surgery (greater than 6 months prior to abrasion)
* Diabetes (Patients with even mild diabetic neuropathy can have decreased pain sensation and also delayed corneal epithelial healing)
* Any eye condition that may be deemed to interfere with the conduct of the protocol or outcome measurement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2019-10-24 (Actual); Study Completion 2019-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hyde, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bandage Contact Lens (BCL) Group | Usual Care Group
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study terminated due to change in practice decreasing availability of eligible patients. No participants were enrolled in the Usual Care Group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bandage Contact Lens (BCL) Group | Usual Care Group | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 1 |  | 1
  >=65 years | 0 |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 0
  Male | 1 |  | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 1 |  | 1
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 0 |  | 0
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Score
Description: Measured on scale of 0 being no pain, 5 being moderate pain and 10 being worst pain possible
Time Frame: Baseline, approx. 12-24 hours, approx. 36-48 hours, approx. 1 day, 3 days, and/or 5 days post-discharge
Population: Study terminated due to change in practice decreasing availability of eligible patients. Data was not collected or analyzed.
Arm/Group | Bandage Contact Lens (BCL) Group | Usual Care Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study for a total of approximately 7 days on all participants.
Description: Study terminated due to change in practice decreasing availability of eligible patients. No participants were enrolled in the Usual Care Group.
Arm/Group | Bandage Contact Lens (BCL) Group | Usual Care Group
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

LIMITATIONS AND CAVEATS:
Study terminated due to change in practice decreasing availability of eligible patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2019-01-24): https://cdn.clinicaltrials.gov/large-docs/14/NCT04159714/Prot_001.pdf